CLINICAL TRIAL: NCT06384313
Title: Prevention of Diabetes with a Novel Butyrate-enriched Triglyceride
Brief Title: Butyrate-enriched Triglyceride and Diabetes Prevention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NL86266.068.24
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes; PreDiabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Prediabetic State; Obesity | interventions — Butyrates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- butyrate/hexanoate-enriched triglycerides (Experimental): Oil containing butyrate and hexanoate-enriched triglycerides
  Interventions: Dietary Supplement: butyrate/hexanoate-enriched triglycerides
- placebo (Placebo Comparator): Oil devoid of butyrate and hexanoate but with similar composition as the intervention oil
  Interventions: Dietary Supplement: butyrate/hexanoate-enriched triglycerides

INTERVENTIONS:
Dietary Supplement: butyrate/hexanoate-enriched triglycerides — The oils are consumed two times a day for 24 weeks (six months).

SUMMARY:
A body of animal studies as well as observational studies in humans demonstrated that butyrate is one SCFA that has pronounced positive effects on body weight control, inflammation, and insulin resistance. Even though the SCFA hexanoate is less researched, it has been shown to be involved in anti-inflammatory processes. Of note, acute human studies showed that fibre-induced metabolic improvements are linked to higher SCFA levels in the systemic circulation. It has been shown that a butyrate/hexanoate-enriched triglyceride oil enhanced systemic butyrate and hexanoate concentrations for a prolonged time. Yet, it remains to be determined whether a chronic increase in circulating butyrate and hexanoate concentrations translate into long-term benefits. In this study it is hypothesized that a chronic increase of butyrate/hexanoate in the circulation may improve host metabolism and metabolic health by improving adipose tissue function, reducing systemic lipid overflow and inflammation thereby increasing peripheral insulin sensitivity in individual with overweight/obesity and prediabetes.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Age 20-70 years
* BMI ≥ 28 and < 40 kg/m2
* Weight stable for at least 3 months
* Normal blood pressure (systolic blood pressure 100-140 mmHg, diastolic blood pressure 60-90 mmHg)
* One or more of the following criteria to determine disturbed glucose/insulin homeostasis

  * Fasting glucose 5.6-6.9 mmol/L
  * Two-hour glucose of 7.8-11.1 mmol/L
  * HOMA-IR ≥ 2.2
  * HbA1c (5.7-6.4%)

Exclusion Criteria:

* Diabetes mellitus (type 1 or 2)

  * Cardiovascular disease: including no history or myocardial infarction, heart failure, arrhythmias
  * Pulmonary disease: no history of chronic obstructive pulmonary disease, emphysema, bronchitis, asthma
  * Kidney (e.g. kidney failure) or liver (e.g. cirrhosis, non-alcoholic fatty acid) malfunction
  * Gastrointestinal disease (no inflammatory bowel disease, irritable bowel syndrome or digestive disorders) or a history of abdominal surgery (except appendectomy and cholecystectomy)
  * Autoimmune disease
  * Any other diseases affecting glucose and/or lipid metabolism or use of any medication that influence glucose or fat metabolism and inflammation
  * Ongoing disease or any disease with a life expectancy ≤ 5 years
  * Abuse of products; alcohol (>15 units per week) and drugs, excessive nicotine use defined as >20 cigarettes per week
  * Regular supplementation of pre- or probiotic products, use of pre- or probiotics, antibiotics and laxatives 3 months prior to the start of the study
  * Intensive exercise training more than three hours a week
  * Plan to lose weight or to follow a hypocaloric diet or vegetarian diet
  * Pregnancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Peripheral insulin sensitivity | Before and 6 months after the start of the intervention
  The change of peripheral insulin sensitivity as assessed by a hyperinsulinaemic-euglycemic clamp

SECONDARY OUTCOMES:
hepatic insulin sensitivity | Before and 6 months after the start of the intervention
  The change in hepatic insulin sensitivity as assessed by a hyperinsulinaemic-euglycemic clamp
adipose tissue insulin sensitivity | Before and 6 months after the start of the intervention
  The change in adipose tissue insulin sensitivity as assessed by a hyperinsulinaemic-euglycemic clamp
Energy expenditure (indirect calorimetry) | Before and 6 months after the start of the intervention
  The change in energy expenditure as measured via ventilated hood system
Substrate oxidation (indirect calorimetry) | Before and 6 months after the start of the intervention
  The change in substrate oxidation as measured via ventilated hood system
circulating SCFA | Before and 6 months after the start of the intervention
  The change in concentrations of circulating SCFA
Faecal SCFA | Before and 6 months after the start of the intervention
  The change in concentrations of faecal SCFA
Faecal microbiota composition | Before and 6 months after the start of the intervention
  The change in faecal microbiota composition assessing abundances of bacteria and diversity indices as assessed via 16s rRNA gene
Circulating hormones such as insulin | Before and 6 months after the start of the intervention
  The change in concentrations of circulating hormones in peripheral blood
Circulating metabolites such as glucose | Before and 6 months after the start of the intervention
  The change in concentrations of metabolites in peripheral blood
body composition | Before and 6 months after the start of the intervention
  The change in body composition as assessed using DEXA scans
body weight | Before and 6 months after the start of the intervention
  The change in body weight in kg using a weight scale
Gut permeability | Before and 6 months after the start of the intervention
  The change in gut permeability as assessed using a multi-sugar test

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No